CLINICAL TRIAL: NCT02009696
Title: ProMRI Study of the Entovis Pacemaker System (Phase B)
Status: Completed | Type: Observational
Sponsor: Biotronik, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: G120226 (Phase B)
Record Dates: First submitted 2013-12-09; First posted 2013-12-12 (Estimated); Results first posted 2015-07-10 (Estimated); Last update posted 2015-11-25 (Estimated); Status verified 2015-10

CONDITIONS: Magnetic Resonance Imaging (MRI); Cardiac Pacing
MeSH Terms: interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Pacemaker Therapy: Patients with a ProMRI Pacemaker System
  Interventions: Device: Patients with a ProMRI Pacemaker System; Other: Magnetic Resonance Imaging (MRI) scan

INTERVENTIONS:
Device: Patients with a ProMRI Pacemaker System — Bradycardia Slow Heart Beat
Other: Magnetic Resonance Imaging (MRI) scan — MRI scan of heart/chest or thoracic spine.

SUMMARY:
The objective of the ProMRI Study (Phase B) is to demonstrate the clinical safety of the ProMRI Pacemaker System when used under specific MRI conditions without scan exclusion zone.

ELIGIBILITY:
Inclusion Criteria:

The following initial inclusion criteria must be met for a subject to be enrolled and considered for the MRI-procedure:

* Age greater than 18 years
* Able and willing to complete MRI testing
* Able to provide written informed consent
* Available for follow-up visit at the study site
* Implanted with a pacemaker system consisting only of an Entovis pacemaker (DR-T, SR-T) and one or two Setrox S 53 or Setrox S 60 pacemaker lead(s). (No leads other than Setrox S (53 or 60 cm) leads may be implanted. This includes lead extensions or abandoned leads in the subject.)
* Pacemaker implanted pectorally
* All pacemaker system components implanted, repositioned, or exchanged at least 5 weeks prior to enrollment
* Underling rhythm identifiable during sensing test
* All pacing thresholds are measureable and are less than or equal to 2.0 V @0.4 ms
* Absence of phrenic nerve stimulation at 4.8V @ 1.0 ms
* Pacing impedance is between 200 and 1500 ohm
* Able and willing to use the Cardio Messenger

At the pre-MRI procedure, the following procedure-related criteria must be met for the subject to undergo the MRI scan:

* Absence of phrenic nerve stimulation at 4.8V @ 1.0 ms

  •|pacing threshold at Pre-MRI follow-up - pacing threshold at baseline| ≤ 0.5 V
* All pacing thresholds are measureable and are ≤ 2.0 V @ 0.4 ms
* The pacemaker system has been implanted for at least 6 weeks.
* Subject did not have a pacemaker or lead explant, exchange or reposition in the previous 6 weeks.
* All lead impedances are between 200 and 1500 ohm.
* Battery status is at least 30% of capacity

Exclusion Criteria:

* Enrolled in any other clinical study
* For pacemaker systems that include an atrial lead, subjects with either

  * Persistent atrial arrhythmia (lasting longer than 7 days or requiring cardioversion)
  * Permanent atrial arrhythmia
* Life expectancy of less than three months
* Pregnancy
* Cardiac surgery expected in the next three months

Implanted with other medical devices that may interact with MRI, such as:

* abandoned pacemaker/ICD leads
* lead extensions
* mechanical valves
* other active medical devices
* non-MRI compatible devices
* other metallic artifacts/components in body that may interact with MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients selected for participation should be from the investigators' general patient population according to the inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 221 (Actual)
Dates: Start 2013-12; Primary Completion 2014-11 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (31):
- United States (31):
  - Phoenix, Arizona
  - Scottsdale, Arizona
  - Concord, California
  - Newport Beach, California
  - Rancho Mirage, California
  - New Haven, Connecticut
  - Newark, Delaware
  - Washington D.C., District of Columbia
  - Valparaiso, Indiana
  - Iowa City, Iowa
  - Lafayette, Louisiana
  - Cumberland, Maryland
  - Boston, Massachusetts
  - Burlington, Massachusetts
  - Worcester, Massachusetts
  - Ann Arbor, Michigan
  - Ypsilanti, Michigan
  - Kansas City, Missouri
  - St Louis, Missouri
  - Flushing, New York
  - New York, New York
  - The Bronx, New York
  - Winston-Salem, North Carolina
  - Toledo, Ohio
  - Salem, Oregon
  - Newtown, Pennsylvania
  - Greenville, South Carolina
  - Amarillo, Texas
  - Mechanicsville, Virginia
  - Virginia Beach, Virginia
  - Spokane, Washington

REFERENCES:
- [Result] Bailey WM, Mazur A, McCotter C, Woodard PK, Rosenthal L, Johnson W, Mela T; ProMRI Study Investigators. Clinical safety of the ProMRI pacemaker system in patients subjected to thoracic spine and cardiac 1.5-T magnetic resonance imaging scanning conditions. Heart Rhythm. 2016 Feb;13(2):464-71. doi: 10.1016/j.hrthm.2015.09.021. Epub 2015 Sep 25. PMID 26409098

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pacemaker Therapy
Started | 221
Completed | 219
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Pacemaker Therapy
Number analyzed (Participants) | 221
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.4 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 82
  Male | 139

OUTCOME MEASURES:

1. Primary Outcome: MRI and Pacing System Related Serious Adverse Device Effect (SADE) Free Rate
Time Frame: 1 Month Post-MRI
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pacemaker Therapy
Number analyzed (Participants) | 221
percentage of participants | 99.5 [97.5 to 100]

2. Primary Outcome: Percentage of Participants Free of Atrial Pacing Threshold Rise
Description: Evaluate the percentage of atrial pacing leads with a pacing threshold increaess between the Pre-MRI and one-month post-MRI follow-up.
Time Frame: Between Pre-MRI and 1 Month Post-MRI
Population: Number of participants with an atrial lead and same atrial threshold polarity (either uni- or bi-polar) at pre-MRI and one-month post-MRI.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pacemaker Therapy
Number analyzed (Participants) | 194
percentage of participants | 100 [98.1 to 100]

3. Primary Outcome: Percentage of Participants Free of Ventricular Pacing Threshold Rise
Description: Evaluate the percentage of ventricular pacing leads with a pacing threshold increase between the Pre-MRI and one-month post-MRI follow-up.
Time Frame: Between Pre-MRI and 1 Month Post-MRI
Population: Number of participants with a ventricular lead and same ventricular threshold polarity (either uni- or bi-polar) at pre-MRI and one-month post-MRI.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pacemaker Therapy
Number analyzed (Participants) | 206
percentage of participants | 100 [98.2 to 100]

4. Primary Outcome: Percentage of Participants Free of P-wave Sensing Attenuation
Description: Evaluate the percentage of subjects who experience P-wave attenuation between the pre-MRI and one-month post-MRI follow-up.
Time Frame: Between Pre-MRI and 1 Month Post-MRI
Population: Number of participants with an atrial lead and same sensing polarity (either uni- or bi-polar) at pre-MRI and one-month post-MRI.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pacemaker Therapy
Number analyzed (Participants) | 170
percentage of participants | 98.2 [94.9 to 99.6]

5. Primary Outcome: Percentage of Participants Free of R-wave Sensing Attenuation
Description: Evaluate the percentage of subjects who experience R-wave attenuation between the pre-MRI and one-month post-MRI follow-up.
Time Frame: Between Pre-MRI and 1 Month Post-MRI
Population: Number of participants with a ventricular lead and same ventricular sensing polarity (either uni- or bi-polar) at pre-MRI and one-month post-MRI.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pacemaker Therapy
Number analyzed (Participants) | 188
percentage of participants | 100 [98.1 to 100]

ADVERSE EVENTS:
Arm/Group | Pacemaker Therapy
Serious Adverse Events (participants affected / at risk) | 22/221
Other Adverse Events (participants affected / at risk) | 38/221
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pacemaker Therapy (N=221)
Angina (Cardiac disorders) | 3 (3)
Arrhythmia (Cardiac disorders) | 3 (3)
Cancer (General disorders) | 1 (1)
Coronary Artery Disease (Cardiac disorders) | 2 (2)
Gastrointestinal (Gastrointestinal disorders) | 2 (2)
Infection (General disorders) | 1 (1)
Medication Related (General disorders) | 1 (1)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 3 (3)
Peripheral Vascular Disease (Vascular disorders) | 1 (1)
Syncope/Pre-Syncope (Cardiac disorders) | 1 (1)
Worsening Chronic Heart Failure (Cardiac disorders) | 1 (1)
General Disorders (General disorders) | 6 (7)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pacemaker Therapy (N=221)
MRI Incidental Finding (General disorders) | 38 (41)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigators agree to submit copies of any manuscript proposed for publication to Sponsor for review at least 30 days in advance of submission for publication or presentation. Sponsor may extend such review period for another 90 days to file patent applications or take other steps to protect its intellectual property interests, or to remove from the paper or presentation any language that is detrimental to Sponsor's intellectual property interests.